CLINICAL TRIAL: NCT05741047
Title: Comparing the Effect of Powdered Skim Milk Containing A2 β-casein Only Versus Conventional Powdered Skim Milk Containing A1 and A2 β-caseins on Mild Cognitive Impairment in Older Adults: a Double-blind, Randomized, Controlled Trial
Brief Title: Comparative Effects of a2 Skim Milk on Mild Cognitive Impairment in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Collaborators: Edanz Group Japan Ltd (Unknown); Beijing Esmile Technology Co. Ltd. (Unknown); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: A2MC-G190549358
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment; Adults
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a2 Group (Active Comparator): The group consuming a2Milk skim milk powder (1L) containing A2 β-casein only
  Interventions: Other: a2Milk skim milk powder
- Control Group (Placebo Comparator): The group consuming Yili skim milk powder (1L) containing A1 and A2 β-caseins
  Interventions: Other: Yili skim milk powder

INTERVENTIONS:
Other: a2Milk skim milk powder — a2Milk skim milk powder (1L) containing A2 β-casein only
  Other Names: Treatment group
  Arms: a2 Group
Other: Yili skim milk powder — Yili skim milk powder (1L) containing A1 and A2 β-caseins
  Other Names: Control group
  Arms: Control Group

SUMMARY:
The aim of the study is to compare the effects of powdered skim milk containing A2 β-casein only versus conventional powdered skim milk containing A1 and A2 β-casein milk on cognition, inflammation, and dietary intake in adults aged 65-75 years.

ELIGIBILITY:
For inclusion in the study, participants must meet all of the following criteria:

1. Adults aged 65-75 years;
2. Complaint of memory loss for more than 6 months;
3. Base on the Chinese version of Mini Mental State Examination (MMSE), cognitive ability score is lower than the standard cut-off value according to age and education levels: MMSE score≤ 17 points if years of education is 0 year; ≤ 20 points if 6 years or less of education; ≤ 24 points if more than 6 years of education
4. Living and social functions are reduced: activities of daily living (ADL) score ≤18;
5. Not meeting the diagnostic criteria for dementia (Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition), Alzheimer Disease (National Stroke Institute for Neuropathic Speech Disorders and Association for Alzheimer Disease and Related Disorders); no mental disorder, brain damage, or other physical disorders that can lead to cognitive impairment.
6. Agreed not to participate in another interventional clinical research study during the present study;
7. Signed informed consent

Participants must be excluded from the study if they meet any of the following criteria:

1. <65 years; or >75 years
2. Neurological examination showed focal signs of central nervous system disorder such as hemiplegia, dysesthesia, aphasia; history of cerebrovascular diseases (including hemorrhagic and ischemic types), internal brain trauma or fracture;
3. Asthmatic bronchitis, severe hypertension, angina and severe infection;
4. Mental disorders such as depression and anxiety; endocrine system diseases (such as hyperthyroidism, hypothyroidism, systemic lupus erythematosus, rheumatoid arthritis);
5. Newly diagnosed, progressing or advanced tumors;
6. Visual, reading, hearing impairment or language communication difficulties that significantly affect cognitive function tests;
7. History of alcohol dependence and abuse of psychoactive substances (e.g., antipsychotics, benzodiazepines, cholinesterase inhibitors, sedatives), or use of drugs that affect cognitive function;
8. Neurological diseases (e.g. Parkinson's disease, epilepsy);
9. Antibiotic treatment in previous 2 weeks;
10. Administered immunosuppressive drugs in the 4-weeks preceding screening;
11. Allergy to milk or dairy;
12. Diagnosed lactose intolerance;
13. Other diseases that investigators judged as unsuitable to participate the study.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Changes of Subtle Cognitive Impairment Test (SCIT) at Visit 2 and Visit 4 compared to baseline | Visit 2 (14 days after baseline); Visit 4 (90 days after baseline); baseline (14 days after enrolment)
  Record responding time and speed on the SCIT test
Changes of serum glutathione (GSH) at Visit 2 and Visit 4 compared to baseline | Visit 2 (14 days after baseline); Visit 4 (90 days after baseline); baseline (14 days after enrolment)
  Record serum glutathione (GSH) (µmol/L) as an anti-oxidation marker

SECONDARY OUTCOMES:
Changes of short-chain fatty acids at Visit 2, 3, and 4 compared to baseline | Visit 2 (14 days after baseline); Visit 3 (28 days after baseline); Visit 4 (90 days after baseline); baseline (14 days after enrolment)
  Record short-chain fatty acids (mg/g) as a faecal marker of inflammation
Changes of quality of life at Visit 4 compared to baseline | Visit 4 (90 days after baseline); baseline (14 days after enrolment)
  Record Healthy Brain Ageing - Functional Assessment Questionnaire via patient self-report as a quality of life measure
Changes of C-reactive protein at Visit 2 and 4 compared to baseline | Visit 2 (14 days after baseline); Visit 4 (90 days after baseline); baseline (14 days after enrolment)
  Record C-reactive protein (mg/L) as a blood marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Keming Zhang, MD, Principal Investigator — The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - General Hospital of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin

REFERENCES:
- [Derived] Zhang K, Sun J, Han M, Diao Y, Xia Y, Yang C, Robinson SR. Milk free of A1 beta-casein supports superior gains in cognition and quality of life, relative to conventional milk, in older adults with mild cognitive impairment. J Nutr Health Aging. 2025 Jul;29(7):100579. doi: 10.1016/j.jnha.2025.100579. Epub 2025 May 14. PMID 40373392